CLINICAL TRIAL: NCT06728709
Title: Lung Assessment and Monitoring in Critically Ill Obstetrics and Gynecological Patients by Point of Care Ultrasound; Prospective Observational Study
Brief Title: Lung Ultrasound in Critically Ill Obstetrics and Gynecological Patients
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU R148/2024
Record Dates: First submitted 2024-08-01; First posted 2024-12-11 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-01

CONDITIONS: Obstetric Complication; Gynecologic Cancer; Lung Diseases; Ultrasound
Keywords: lung ultrasound; critically ill peripartum; critically ill gynecological cases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obstetrics critically ill: critically ill obstetrics patients admitted yo ICU for any cause during pregnancy or postpartum.
  Interventions: Diagnostic Test: ultrasound detection of any abnormal ultrasonographical findings.
- gynecological critically ill patients: gynecological cases admitted to ICU for any cause of medical or postoperative care
  Interventions: Diagnostic Test: ultrasound detection of any abnormal ultrasonographical findings.

INTERVENTIONS:
Diagnostic Test: ultrasound detection of any abnormal ultrasonographical findings. — ultrasound assessment within 24 hours. Then reassessment every 48 hours or when the patient develops respiratory distress.
  While the patient is in a supine or semi-recumbent position, and the probe is in a short axis. The 8-region technique will be used. The areas are four on each side of the chest. The examiner will assess 8 regions -Anterior chest wall ( ACW), Anterior axillary line (AAXL), costo-phrenic angle (COSTO), Postero-lateral alveolar &/ or pleural syndrome (PLAPS) right and left . Each region will be scored using the LUS aeration score. as follows: "0," A-pattern with 0-2 B-lines; "1," more than 2 separated B-lines; "2," multiple coalescent B-lines; or "3," lung consolidation, . A global LUS score will be calculated at each time point and range from 0 to 24.
  posterior region will be assessed if needed and if feasible. The venous status will be assessed through a subcostal view for inferior vena cava diameter.

SUMMARY:
Pulmonary dysfunction aggravates the illness of critically ill obstetrics and gynecological patients. Early identification with bedside technique and prompt management may improve the outcome of critical care in this vulnerable population

DETAILED DESCRIPTION:
Hormonal changes in a woman's menstrual cycle and changes during pregnancy affect the respiratory system. These changes especially during pregnancy and peripartum complicate the critical care management of the female patients. In addition to the effect of different pregnancy-related as sepsis, and preeclampsia which directly or indirectly predispose to pulmonary complications.

The presence of difficulty in the transfer of critically ill patients mandates point of care modality. Avoidance of fetal exposure to hazardous radiation demands safe technology. Ultrasound arises as a screening method that can be performed rapidly and enables healthcare providers to make timely decisions with no radiation exposure. Thus it facilitates the management of critically ill obstetric and gynecological patients.

When compared to other imaging techniques; X-ray imaging is preferably restricted in parturient because of the ionizing risk on the fetus, and CT is not feasible in critically ill if there is a risk of transfer. Thus ultrasound emerged as a bedside imaging technique.

Yet, the prevalence of the specific ultrasound signatures in that population is not clearly defined and its relation to poor outcome was not tested, This trial is the first trial to determine frequency, timing concerning admission, type of pulmonary abnormalities detectable by LUS, and their associations with poor outcome in patients whether obstetrics or gynecology admitted to the ICU specialized in women's intensive care

ELIGIBILITY:
Inclusion Criteria:

* Any patient admitted to the obstetrics and gynecology intensive care unit

Exclusion Criteria:

* Patient's refusal
* inability to do a lung ultrasound examination during the first 24 hours of admission

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant, peripartum, or gynecological critical illness
Study Population: critically ill women admitted in the ICU for any medical, obstetric, or surgical causes.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
the Prevalence of different ultrasonographical abnormal lung signatures | From date of admission untill Death from any cause or discharge from ICU, whichever comes first. assessed up to 20 days
  presence or absence of us abnormalities as: abnormal sliding, interstitial syndrome, consolidation, cavitation, pleural effusion, or collapse

SECONDARY OUTCOMES:
correlation of ultrasonographic finding with mortality or poor outcome | from the appearance of abnormal ultrasonographic signature to death or disharge from ICU which comes first , assessed up to 20 days from the day of admission
  frequency of occurrence of poor outcomes -mortality or ventilatory support- for every abnormal lung ultrasonographic signature.
timing of appearance of abnormal ultrasonography lung signatures | on admission, after every 48 hours during ICU stay till death or dischrage from ICU which comes first, assessed up to 20 days from admission
  the time of detection of the abnormal lung ultrasonographic finding

CONTACTS AND LOCATIONS:
Overall Officials: wessam selima, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rocca E, Zanza C, Longhitano Y, Piccolella F, Romenskaya T, Racca F, Savioli G, Saviano A, Piccioni A, Mongodi S. Lung Ultrasound in Critical Care and Emergency Medicine: Clinical Review. Adv Respir Med. 2023 May 17;91(3):203-223. doi: 10.3390/arm91030017. PMID 37218800
- [Background] Pisani L, De Nicolo A, Schiavone M, Adeniji AO, De Palma A, Di Gennaro F, Emuveyan EE, Grasso S, Henwood PC, Koroma AP, Leopold S, Marotta C, Marulli G, Putoto G, Pisani E, Russel J, Serpa Neto A, Dondorp AM, Hanciles E, Koroma MM, Schultz MJ. Lung Ultrasound for Detection of Pulmonary Complications in Critically Ill Obstetric Patients in a Resource-Limited Setting. Am J Trop Med Hyg. 2020 Dec 14;104(2):478-486. doi: 10.4269/ajtmh.20-0996. PMID 33319731